CLINICAL TRIAL: NCT04471467
Title: Effect of Tracheal Tube Fixation Method on Nasal Pressure of Patients With Nasal Tracheal Intubation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yu Sun, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: PUs
Record Dates: First submitted 2020-07-12; First posted 2020-07-15 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Nasotracheal Intubation
Keywords: nasotracheal intubation; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group F: Using tracheal tube fixation method （According to the needs of the surgery, the surgeon who did not participate in the trial）
  Interventions: Procedure: Fixed tracheal tube
- group N: No tracheal tube fixation （According to the needs of the surgery, the surgeon who did not participate in the trial）

INTERVENTIONS:
Procedure: Fixed tracheal tube — Tracheal tube fixation is determined by the surgeon according to the needs of the operation and is an independent process. Our research simply installed a monitoring device between the tube and the nose. The tube fixation takes place whether the observation of pressures is agreed to or not, as per standard protocol.
  Groups: group F

SUMMARY:
Nasotracheal intubation (NTI) is commonly used in operations of the mouth, pharynx, larynx and also the neck .Various complications can occur such as epistaxis, bacteremia,turbinectomy, retropharyngeal dissection, and nasal alar pressure sores or necrosis.In clinical practice, nasal pressure sores caused by NTI are not uncommon, but have failed to attract clinical attention.The investigators have observed that the surgeon fixed the nasal tracheal tube and threaded tube directly to the patient's head. The investigators suspect that this method can reduce the pressure between the nasal tube and the nose.

DETAILED DESCRIPTION:
Nasotracheal intubation (NTI) is commonly used in operations of the mouth, pharynx, larynx and also the neck .Various complications can occur such as epistaxis, bacteremia,turbinectomy, retropharyngeal dissection, and nasal alar pressure sores or necrosis.In clinical practice, nasal pressure sores caused by NTI are not uncommon, but have failed to attract clinical attention.Oral and maxillofacial surgery usually uses nasal endotracheal intubation to manage the airway. The tube fixation directly presses the skin of the patient's nose. Due to the operation, the surgeon must stand on the head of the patient and there is not enough space to place the tracheal tube bracket. Prolonged vascular compression on the nasal region may be caused by excessive tension and angulation of the nasotracheal tube against the nasal tissue.Studies have proposed the use of nasal packing, hydrocolloidal dressing and modified nasal tracheal tube to reduce the direct contact between the nasal tube and the nose, relieve the pressure between the two, so as to prevent the occurrence of alar pressure ulcers, but there is no objective data to show the degree of pressure reduction.In clinical practice, the investigatorshave observed surgeons fixed the nasal endotracheal tube and threaded the tube directly to the patient's head. The investigators suspect that this method can reduce the pressure between the nasal tube and the nose, so the investigators want to use a pressure sensor to monitor the pressure between the two.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years old
* ASA physical status I and II
* Requiring general anesthesia with nasal intubation

Exclusion Criteria:

* Previous history of pressure ulcers
* Nasal trauma or defect
* The need for emergency surgery
* Contraindications to nasal intubation
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who will be receiving general anesthesia with nasal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
pressure between the nasal tube and nose | Immediately after procedure
  pressure between the nasal tube and nose under different conditions